CLINICAL TRIAL: NCT06686199
Title: Potato Diet Intervention Study in a College Population
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yu Zhang (Other)
Responsible Party: Sponsor-Investigator, Yu Zhang, professor, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT_ Potato Meal
Record Dates: First submitted 2024-07-15; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-07

CONDITIONS: Metabolism and Nutrition Disorder
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator)
  Interventions: Dietary Supplement: steamed potato
- Intervention group (Experimental)
  Interventions: Dietary Supplement: fried potato

INTERVENTIONS:
Dietary Supplement: steamed potato — 135 g per day 4-5 times per week for 8 weeks
  Arms: Control group
Dietary Supplement: fried potato — 135 g per day 4-5 times per week for 8 weeks
  Arms: Intervention group

SUMMARY:
The goal of this study is to investigate the effects of a potato-based diet intervention on Chinese university students. Employing a randomized controlled double-blind trial design, the intervention will span 8 weeks. The primary objectives include:

* Examining the impact of the potato-based diet intervention on the overall glucose and lipid metabolism levels of university students;
* Exploring the interactions between the potato-based diet intervention and individual metabolic profiles and glucose-lipid metabolic pathways;
* Analyzing the association between the potato-based diet intervention and gut health through gut microbiota analysis.

Participants will undergo either the potato-based diet intervention or the control group treatment. Changes in waist circumference, blood pressure, blood glucose, and blood lipid levels will be observed to assess the effects of the potato-based diet on university students' health. Additionally, alterations in metabolic profiles and glucose-lipid metabolic pathways will be analyzed, along with gut microbiota analysis, to investigate the relationship between the potato-based diet and gut health.

DETAILED DESCRIPTION:
This study aims to recruit young adults aged 18-35 from university populations who meet the criteria and are willing to participate. After screening based on baseline information, eligible volunteers will be randomly assigned to two groups: an intervention group and a control group. The intervention group will consume fried potatoes, while the control group will consume steamed potatoes, at a daily dose of 135g, 4-5 times a week, for an 8-week dietary intervention period.

1. The effects of potato-based dietary intervention on the metabolic profiles of glucose and lipids in the human body will be assessed. General indicators such as height, weight, blood pressure, waist circumference, and hip circumference will be measured at baseline and at the intervention endpoint for all participants. Fasting blood samples will be collected to measure four lipid parameters (TG, TC, LDL-C, HDL-C), fasting blood glucose, fasting insulin, glycosylated hemoglobin levels, and serum C-peptide levels. Changes and differences in glucose and lipid metabolism indicators among groups will be observed.
2. The role of potato-based dietary intervention on the blood metabolic profiles, gut microbiota composition, and inflammatory response in university student populations will be investigated. Blood and stool samples will be collected to study the effects of potato-based dietary intervention on metabolic markers of glucose and lipids in biological samples and the gut microbiota composition in fecal samples. The analysis will focus on its effects on serum inflammatory factors by influencing glucose and lipid metabolism pathways and gut microbiota composition, as well as inflammatory signaling pathways, elucidating the mechanisms through which it modulates glucose and lipid metabolism.

ELIGIBILITY:
Inclusion Criteria:

* University students at school

Exclusion Criteria:

* Smoking (≥1 cigarette/week);
* heavy alcohol consumption (>224 g/week for men and >168 g/week for women);
* diabetes, heart disease, stroke, high blood pressure, liver dysfunction, kidney dysfunction, or gastrointestinal disorders;
* taking dietary supplements (e.g., vitamins, minerals, probiotics, or prebiotics);
* taking medications (e.g., aspirin, statin, or antihypertensive medications);
* within the past 3 months taken antibiotics;
* had surgery in the past 3 months;
* participated in other clinical studies in the past 3 months;
* preference for fried and baked foods.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in body weight from baseline | Time Frame: 2 months
  The investigators will measure body weight before and after treatment.
Change in blood glucose from baseline | Time Frame: 2 months
  The investigators will measure fasting plasma glucose levels in blood samples before and after treatment.
Change in triglycerides from baseline | 2 month
  The investigators will measure Triglyceride levels in blood samples before and after treatment.

SECONDARY OUTCOMES:
Change in lipid indicators from baseline | 2 month
  The investigators will measure total cholesterol, LDL-C, and HDL-C levels in blood samples before and after treatment.

IPD SHARING:
Plan to Share IPD: No